CLINICAL TRIAL: NCT00089271
Title: A Phase I Study Of 17-Dimethylaminoethylamino-17-Demethoxygeldanamycin, (17-DMAG) (NSC 707545) In Patients With Advanced Solid Tumors
Brief Title: 17-DMAG in Treating Patients With Metastatic or Unresectable Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02620; PCI-03-153; U01CA069912 (NIH); U01CA099168 (NIH); U01CA062502 (NIH); CDR0000378189 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — 17-(dimethylaminoethylamino)-17-demethoxygeldanamycin

ARMS (1):
- Treatment (alvespimycin hydrochloride) (Experimental): Patients receive 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG) IV over 1-6 hours on days 1-3 or 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alvespimycin hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: alvespimycin hydrochloride — Given IV
  Other Names: 17-DMAG HCL; KOS-1022
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of 17-DMAG in treating patients with metastatic or unresectable solid tumors or lymphomas. Drugs used in chemotherapy, such as 17-DMAG, work in different ways to stop cancer cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG) in patients with metastatic or unresectable solid tumors or lymphomas.

II. Determine the safety and toxicity of this drug in these patients. III. Determine the pharmacokinetics and pharmacodynamics of this drug in these patients.

IV. Determine the recommended phase II dose of this drug for future studies.

SECONDARY OBJECTIVES:

I. Determine tumor response in patients treated with this drug.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG) IV over 1-6 hours on days 1-3 or 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 1-2 patients receive accelerated escalating doses of 17-DMAG until at least 1 of 2 patients experience dose-limiting toxicity (DLT). Cohorts are then expanded to 3-6 patients who receive escalating doses (in a standard manner) of 17-DMAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT.

Patients are followed at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor or lymphoma

  * Metastatic or unresectable disease
* Standard curative or palliative measures do not exist or are no longer effective
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* ALT and AST ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ normal
* Creatinine ≤ 1.25 times ULN
* Creatinine clearance ≥ 60 mL/min
* QTc < 450 msec for male patients (470 msec for female patients)
* LVEF > 40% by MUGA
* No history of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No myocardial infarction or active ischemic heart disease within the past year
* No New York Heart Association class III or IV congestive heart failure
* No poorly controlled angina
* No uncontrolled dysrhythmia requiring medication
* No left bundle branch block
* No history of congenital long QT syndrome
* No other significant cardiac disease
* Pulse oximetry at rest or on exercise > 88%
* No symptomatic pulmonary disease (e.g., chronic obstructive or restrictive pulmonary disease, etc.) or any of the following are allowed:

  * Pulmonary disease requiring medication
  * History of dyspnea, dyspnea on exertion, or paroxysmal nocturnal dyspnea
  * Patients meeting the Medicare criteria for home oxygen or are on oxygen
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double barrier contraception 1 week before, during, and for at least 2 weeks after study participation
* No uncontrolled illness
* No active or ongoing infection
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG)
* No psychiatric illness or social situation that would preclude study compliance
* No concurrent routine colony-stimulating factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Concurrent hormonal therapy allowed
* At least 4 weeks since prior radiotherapy and recovered
* No prior radiation that included the heart in the field (e.g., mantle)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents or therapies
* No concurrent medication that would prolong the QTc interval
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-07; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of alvespimycin hydrochloride | 21 days
Toxicity graded using the NCI CTCAE version 3.0 | Up to 4 weeks
Recommended phase II dose (RP2D) of alvespimycin hydrochloride for future studies determined by toxicity assessments | 21 days
Pharmacokinetics of alvespimycin hydrochloride in blood, urine, and tumor tissue | 21 days
  Analyzed by both non-compartmental and compartmental methods.

SECONDARY OUTCOMES:
Tumor response assessed by tumor measurements | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Belani, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States